CLINICAL TRIAL: NCT04598568
Title: Post-market Clinical Follow-up on the balanSys UNI Knee Prosthesis Implanted With a Spacer Block Surgical Technique
Status: Completed | Type: Observational
Sponsor: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140206_Protocol_V5
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- balanSys UNI knee prosthesis: Participants treated with a balanSys® UNI knee prosthesis
  Interventions: Device: balanSys UNI

INTERVENTIONS:
Device: balanSys UNI — Implantation of a balanSys UNI knee prosthesis implanted with a spacer block surgical technique

SUMMARY:
The purpose of the study is the evaluation of the clinical and radiological long-term performance of the balanSys UNI fix in a multicenter routine clinical setting.

DETAILED DESCRIPTION:
Prospective multicenter follow-up study which examines the short- to long-term post-market clinical data on the safety and performance of the balanSys UNI fix knee prosthesis.

In total at least 100 participants in 3 clinics are included in this multicenter study.

The primary endpoint of the study is the Knee Society Score (KSS) 2 years after surgery.

The following parameters will be collected during the regular clinical and radiological follow-up: Knee Society Score, Knee and Osteoarthritis Outcome Score (KOOS), radiographic evaluation and detection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (signed by participant and investigator)
* Primary implantation
* Age at inclusion: Between 18 and 90 years old
* Willing to participate in the follow-up

Exclusion Criteria:

* Missing Informed consent form
* Known or suspected non-compliance (e.g. drug or alcohol abuse)
* Enrollment of the investigator, his/her family, employees and other dependent persons
* Patient younger than 18 years old
* Revision surgery
* Does have a known allergy to metal in medical devices
* Suffers from ACL rupture
* Pregnancy or in the breast feeding period

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: according to Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 2 years
  The primary endpoint of the study is the Knee Society Score (KSS) 2 years after surgery
  The Knee Society Score consists of an objective score (0-100 points) and a score for function (0-100 points).
  A higher score means a better outcome.

SECONDARY OUTCOMES:
Radiographic evaluation of lucent lines | 6-12 weeks - 10 years
  The second endpoint of interest is the incidence of lucent lines measured in millimeters by means of standard X-rays.
Adverse Events and Complications | 6-12 weeks - 10 years
  Documentation of complication(s):
  - Description of complication with the UKA
  Documentation of component revision(s) (Adverse Events):
  * Reason(s) for revision(s)
  * Revised component(s)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tille E, Beyer F, Auerbach K, Tinius M, Lutzner J. Better short-term function after unicompartmental compared to total knee arthroplasty. BMC Musculoskelet Disord. 2021 Apr 2;22(1):326. doi: 10.1186/s12891-021-04185-w. PMID 33810795